CLINICAL TRIAL: NCT06100484
Title: Potential Impact of Blood Pressure Variability on Right Ventricular Remodeling in Pregnant Women With Pre-eclampsia or Gestational Hypertension
Brief Title: Blood Pressure Variability Effect on Right Ventricular Strain in Women With Hypertensive Disorders With Pregnancy
Status: Completed | Type: Observational
Sponsor: Aswan University (Other)
Responsible Party: Principal Investigator, Mahmoud Elsayed Abdellatif, Cardiology resident, Aswan University
Other Study IDs: RV strain and PET
Record Dates: First submitted 2023-10-20; First posted 2023-10-25 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Hypertension, Pregnancy Induced; Preeclampsia
Keywords: Blood; Pressure; Variabilty; Gestational hypertension; Pre-eclampsia
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Pre-Eclampsia | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy group: Pregnant women above 20 weeks of pregnancy with no hypertensive disorders with pregnancy
  Interventions: Diagnostic Test: Echocardiography
- Diseased group: Pregnant women above 20 weeks of pregnancy with gestational hypertension or pre-eclampsia
  Interventions: Diagnostic Test: Echocardiography

INTERVENTIONS:
Diagnostic Test: Echocardiography — Two-dimensional RV strain imaging will be performed by using three consecutive cardiac cycles of 2D images in the apical four-chamber view to assess RV-GLS

SUMMARY:
The goal of this observational study is to learn about the potential effect of blood pressure variability changes on right ventricular strain in pregnant women with gestational hypertension or pre-eclampsia

DETAILED DESCRIPTION:
Hypertensive disorders of pregnancy include chronic hypertension, gestational hypertension, pre-eclampsia and chronic hypertension with superimposed pre-eclampsia. Pre-eclampsia, and all hypertensive disorders affect about 5-10% of pregnancies.

The term Blood Pressure Variability is an entity that characterizes the continuous and dynamic fluctuations that occur in blood pressure levels throughout a lifetime.

It encompasses a wide range of blood pressure variations; occurring over seconds or minutes (very short- term BPV), along 24 hours (short- term BPV, usually assessed by ambulatory BP monitoring), and between days (mid- term or day- to- day BPV, assessed with home BP monitoring), Long-term BPV has also been described, including seasonal BP variations and changes between clinic visits over months or years (visit- to- visit BPV).

Studies showed that visit-to-visit BP variability was associated with gestational hypertension and preeclampsia , as well as with risk of adverse birth outcomes in pregnant women without proteinuria or chronic hypertension.

Preeclampsia is a pregnancy-specific disorder that complicates 2-8% of pregnancies worldwide.

Traditionally the condition is diagnosed in the case of de novo development of hypertension (> 140/90 mmHg) and proteinuria during the second half of pregnancy (>20 weeks of gestation).

Preeclampsia (PE) is a life-threatening condition in pregnancy and a major cause of maternal and neonatal morbidity and mortality.

It affects 2-8% of pregnancies that develop serious complications such as eclampsia, hemolysis, elevated liver enzyme levels,thrombocytopenia, and pulmonary edema. These end organ damages usually disappear 12 weeks after delivery.

Gestational hypertension refers to hypertension with onset in the latter part of pregnancy (>20 weeks' gestation) without any other features of preeclampsia, and followed by normalization of the blood pressure postpartum, however, be a harbinger of chronic hypertension later in life as compared with patients who do not have such a history.

There is an association between RV longitudinal strain and functional capacity in hypertensive patients. as well as the strong relationship between RV longitudinal strain and cardiovascular mortality and morbidity in a wide range of cardiovascular conditions.

Over the past few decades, there has been a lot of research done on left ventricular remodeling in hypertensive diseases of pregnancy, especially in gestational hypertension and preeclampsia.However, anatomical, functional, and mechanical changes to the right ventricle are still largely unclear. The limited data are also contradictory because some authors reported significant functional changes in the form of increased RV diameter, elevated pulmonary pressure, and decreased RV longitudinal strain. while other studies showed no difference in RV structure and function between normotensive controls and pregnant women with hypertensive disorders.

In the current study, we are going to assess the impact of gestational hypertension and preeclampsia on RV remodeling. If remodeling occurs, we are going to assess RV recovery post partum.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ages equal to or more than 18 years old.
* women with gestational hypertension ( systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg after 20 weeks of gestation without proteinuria ).
* Women with pre-eclampsia (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg after 20 weeks of gestation with proteinuria < 300mg /24 h).

Exclusion Criteria:

* Pregnancy less than 20 weeks gestation.
* Patients with congenital heart diseases.
* Patients with moderate to severe valvular heart diseases.
* Patients with cardiomyopathy whatever its cause.
* Patients with underlying right ventricular dysfunction.
* Poor image quality.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women after 20 weeks of pregnancy
Study Population: Pregnant women after 20 weeks of pregnancy
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-10-06 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Number of participants that experienced right ventricular remodeling | From Baseline at time of examination till 3 months post-partum
  Assessment of right ventricular strain via 2D Echocardiography and Speckle tracking

CONTACTS AND LOCATIONS:
Locations (1):
- Mahmoud Elsayed Abdellatif, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Hutcheon JA, Lisonkova S, Joseph KS. Epidemiology of pre-eclampsia and the other hypertensive disorders of pregnancy. Best Pract Res Clin Obstet Gynaecol. 2011 Aug;25(4):391-403. doi: 10.1016/j.bpobgyn.2011.01.006. Epub 2011 Feb 18. PMID 21333604
- [Background] Chen SSM, Leeton L, Castro JM, Dennis AT. Myocardial tissue characterisation and detection of myocardial oedema by cardiovascular magnetic resonance in women with pre-eclampsia: a pilot study. Int J Obstet Anesth. 2018 Nov;36:56-65. doi: 10.1016/j.ijoa.2018.07.004. Epub 2018 Aug 2. PMID 30143429
- [Background] Levine LD, Ky B, Chirinos JA, Koshinksi J, Arany Z, Riis V, Elovitz MA, Koelper N, Lewey J. Prospective Evaluation of Cardiovascular Risk 10 Years After a Hypertensive Disorder of Pregnancy. J Am Coll Cardiol. 2022 Jun 21;79(24):2401-2411. doi: 10.1016/j.jacc.2022.03.383. PMID 35710191
- [Background] Liu J, Yang L, Teng H, Cao Y, Wang J, Han B, Tao L, Zhong B, Wang F, Xiao C, Wan Z, Yin J. Visit-to-visit blood pressure variability and risk of adverse birth outcomes in pregnancies in East China. Hypertens Res. 2021 Feb;44(2):239-249. doi: 10.1038/s41440-020-00544-7. Epub 2020 Sep 7. PMID 32895496